CLINICAL TRIAL: NCT06127368
Title: An Open-label, Active-controlled, Parallel and Dose-escalation, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Intramuscular (IM) and Subcutaneous (SC) Donepezil (GB-5001) Injections Versus Donepezil Oral Tablet (Aricept®) in Healthy Male Volunteers
Brief Title: Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics From Single Dose of Intramuscular (IM) and Subcutaneous (SC) Donepezil (GB-5001) Injections Versus Donepezil Oral Tablet (Aricept®) in Healthy Male Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: G2GBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GB5001A101
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Cohort Studies

STUDY DESIGN:
Intervention Model Description: sequential
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GB-5001A (Experimental): GB-5001 Suspension for IM/SC injection at three doses(low, intermediate, high) The cohort is determined through random allocation.
  Interventions: Drug: GB-5001A
- GB-5001D (Experimental): GB-5001 Suspension for SC injection at three doses(low, intermediate, high) The cohort is determined through random allocation.
  Interventions: Drug: GB-5001D
- Oral cohort (Active Comparator): Aricept® tablet. The cohort is determined through random allocation.
  Interventions: Drug: Oral cohort

INTERVENTIONS:
Drug: GB-5001A — Depending on the cohort, volume will be varied to administer, and the dosage and route of administration may be varied.
  Arms: GB-5001A
Drug: GB-5001D — Depending on the cohort, volume will be varied to administer.
  Arms: GB-5001D
Drug: Oral cohort — Single dose of Aricept tablet.
  Arms: Oral cohort

SUMMARY:
This study is to evaluate the safety and tolerability of single dose of GB-5001 (donepezil) IM and SC depot in healthy male Adults. And, It is to evaluate pharmacokinetic characteristics of GB-5001 (donepezil) IM and SC single dose injection vs. active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males,19 to 55 years of age, inclusive at the time of screening visit
* Subject with a body weight of 55 kg or more and a body mass index (BMI) equal to or greater than 18.5 kg/m² but less than 30 kg/m²
* Subject without congenital or chronic conditions, and with no pathological symptoms or findings on internal medical examination
* Subject who has been deemed suitable based on screening test results assessed by the principal investigator
* Subject who can understand this clinical trial, provide informed written consent prior to the clinical trial procedures

Exclusion Criteria:

* Subjects with the following medical history or symptoms, as determined by the Principal Investigator to pose a risk to the trial.

  * Renal/Genitourinary, Gastrointestinal, Cardiovascular, Cerebrovascular, Pulmonary, Endocrine, Immune, Musculoskeletal, Neurological, Psychiatric, Dermatological, and Hematological conditions.
  * Rhabdomyolysis
  * Seizure, Epilepsy, Fainting
  * peptic ulcer or gastrointestinal hemorrhage
  * Gastrointestinal pathology, uncontrollable gastrointestinal symptoms or a history of disturbing absorption, distribution, metabolism or excretion
  * Severe physical/organ abnormalities
  * Human immunodeficiency virus, Hepatitis B virus, Hepatitis C virus
* Subjects with a history of, or currently receiving, the following medications, as determined by the Principal Investigator regarded as a risk to the trial.

  * Medications, including antidepressants, that can induce Rhabdomyolysis
  * Medications with a risk of ulcer development.
  * Potent inhibitors of cytochrome P450 (CYP) enzymes
  * Anticholinergic drugs, cholinomimetics, and other cholinesterase inhibitors
* Subjects who have difficulty with venipuncture or injection procedures via catheter or intravenous access
* Subjects who have been consistently engaging in excessive smoking or consuming caffeine or alcohol within the last 3 months prior to screening, or Subjects who cannot abstain from smoking, caffeine, and alcohol consumption for at least 2 days before the scheduled administration of the investigational product or during the inpatient period

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-01-03 (Estimated); Primary Completion 2024-09-17 (Estimated); Study Completion 2025-01-14 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Part A: Cohort A, B : Upto Day 106 / Cohort C : Upto Day 71 / Cohort D : Upto Day 18, Part B: Cohort E, F, M : Upto Day 18 or Day 106
  Number of participants with adverse events
Clinical Laboratory tests | Part A: Cohort A, B : Upto Day 99 / Cohort C : Upto Day 64 / Cohort D : Upto Day 11, Part B: Cohort E, F, M : Upto Day 64 or Day 99
  Incidence of abnormal clinically significant clinical laboratory test results. (Hematology, Blood Chemistry Test, Urine Test, Blood Coagulation Test, Serum Test and Urine Drug Screening Test.) /Day 1 to Day
Vital Signs | Part A: Cohort A, B : Upto Day 99 / Cohort C : Upto Day 64 / Cohort D : Upto Day 11, Part B: Cohort E, F, M : Upto Day 64 or Day 99
  Incidence of abnormal clinically significant vital signs.(Systolic and Diastolic Blood Pressure, Pulse Rate, Body Temperature)
Physical examination | Part A: Cohort A, B : Upto Day 99 / Cohort C : Upto Day 64 / Cohort D : Upto Day 11, Part B: Cohort E, F, M : Upto Day 64 or Day 99
  Incidence of abnormal clinically significant Physical examination. (This includes an evaluation of the overall appearance and a review of the physical organ systems through questioning, visual inspection, and palpation.)
Electrocardiograms | Part A: Cohort A, B : Upto Day 99 / Cohort C : Upto Day 64 / Cohort D : Upto Day 11, Part B: Cohort E, F, M : Upto Day 64 or Day 99
  Incidence of abnormal clinically significant ECG results (Ventricular rate (beats/min), PR interval (msec), QRS (msec), QT (msec), QTc (msec)

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) | Part A: Cohort A, B : upto Day 99 / Cohort C : upto Day 64 / Cohort D : Upto Day 11 , Part B: Cohort E, F, M : upto Day 11 or Day 99
Pharmacokinetics (Tmax) | Part A: Cohort A, B : upto Day 99 / Cohort C : upto Day 64 / Cohort D : Upto Day 11 , Part B: Cohort E, F, M : upto Day 11 or Day 99
Pharmacokinetics (Tlag) | Part A: Cohort A, B : upto Day 99 / Cohort C : upto Day 64 / Cohort D : Upto Day 11 , Part B: Cohort E, F, M : upto Day 11 or Day 99
Pharmacokinetics (AUCinf) | Part A: Cohort A, B : upto Day 99 / Cohort C : upto Day 64 / Cohort D : Upto Day 11 , Part B: Cohort E, F, M : upto Day 11 or Day 99
Pharmacokinetics (AUClast) | Part A: Cohort A, B : upto Day 99 / Cohort C : upto Day 64 / Cohort D : Upto Day 11 , Part B: Cohort E, F, M : upto Day 11 or Day 99
Pharmacokinetics (AUC 0-762) | Part A: Cohort A, B : upto Day 99 / Cohort C : upto Day 64 / Cohort D : Upto Day 11 , Part B: Cohort E, F, M : upto Day 11 or Day 99
Pharmacokinetics (CL/F) | Part A: Cohort A, B : upto Day 99 / Cohort C : upto Day 64 / Cohort D : Upto Day 11 , Part B: Cohort E, F, M : upto Day 11 or Day 99
Pharmacokinetics (Vd/F) | Part A: Cohort A, B : upto Day 99 / Cohort C : upto Day 64 / Cohort D : Upto Day 11 , Part B: Cohort E, F, M : upto Day 11 or Day 99
Pharmacokinetics (t1/2) | Part A: Cohort A, B : upto Day 99 / Cohort C : upto Day 64 / Cohort D : Upto Day 11 , Part B: Cohort E, F, M : upto Day 11 or Day 99

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea